CLINICAL TRIAL: NCT07285135
Title: Investigating the Effects of Dietary Glycine Supplementation in Patients With Metabolic Dysfunction-associated Steatotic Liver Disease
Brief Title: Dietary Glycine Supplementation in Metabolic Dysfunction-associated Steatotic Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-1240; CSAINV25jan-0007 (Other: NMRC)
Record Dates: First submitted 2025-11-18; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Dysfunction Associated Fatty Liver Disease
Keywords: Fatty liver; Randomized controlled trial; glycine supplements
MeSH Terms: conditions — Fatty Liver | interventions — Glycine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glycine (Active Comparator): 9g per day of glycine in capsules
  Interventions: Dietary Supplement: Glycine
- Placebo (Placebo Comparator): Microcrystalline cellulose in capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glycine — 9g/day of glycine in capsules
  Arms: Glycine
Dietary Supplement: Placebo — Microcrystalline cellulose in identifically-looking capsules
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine whether taking glycine, a naturally occurring amino acid, as a supplement improves liver health measurements in individuals with Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD).

This project will be divided into two parts. The first part will be a case-control study comparing parameters of glycine-dependent metabolic pathways between individuals with MASLD and healthy controls. The second part will be a randomized placebo-controlled trial (RCT) to evaluate the impact of 26-week dietary glycine supplementation on parameters of liver health versus 26-week placebo in patients with MASLD.

DETAILED DESCRIPTION:
This study will recruit 60 participants with MASLD and 30 healthy controls.

Following written informed consent, subjects will be screened. Eligible study subjects will return to undergo MRI scans of the abdomen to measure fat, iron, fibro-inflammation in the liver. Baseline metabolic measurements will include clinical laboratory tests, anthropometrics, body composition, resting energy expenditure, and comprehensive metabolomic profiling. Medical history, physical activity, dietary intake, and sleep quality will also be documented.

Study subjects in with MASLD will be randomized to consume either 9g/day of glycine capsules or placebo capsules for the next 26 ± 4 weeks. Subjects MASLD will be reviewed at 12 ± 4 weeks following the initiation of glycine or placebo to monitor compliance and adverse events.

The final study visit (for subjects with MASLD) will be scheduled at 26 ± 4 weeks after initiation of glycine or placebo. The study subjects will undergo metabolic measurements similar to those performed during the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Age 21-70 years
2. Ability to provide informed consent.

MASLD group:

1. Hepatic steatosis on MRI
2. BMI of 25-50 kg/m2

Controls:

1. Absence of hepatic steatosis on MRI
2. BMI of 18.5-24.9 kg/m2
3. No chronic disease
4. No long-term medications

Exclusion Criteria:

1. Uncontrolled diabetes (HbA1c > 8%)
2. Type 1 Diabetes Mellitus
3. Clinically significant anemia (Haemoglobin < 10 g/dL)
4. Chronic liver disorders (except MASLD) such as Hepatitis B, Hepatitis C, Wilson's disease, hemochromatosis, autoimmune hepatitis, chronic cholestatic disorders, and liver cirrhosis
5. Drugs that may induce hepatic steatosis, such as methotrexate, amiodarone, tamoxifen, or Systemic steroid usage (eg. prednisolone, hydrocortisone, cortisone, dexamethasone)
6. Glomerular filtration rate (GFR < 30 ml/min)
7. Serum alanine transaminase (ALT) > 3x upper limit of normal (ULN)
8. Serum aspartate transaminase (AST) > 3x ULN
9. Liver cirrhosis
10. Significant alcohol consumption (> 20g/day for women and >30g/day for men)
11. Receiving weight loss medications or GLP-1 receptor agonists
12. Pregnancy
13. Uncontrolled thyroid disease
14. Previous bariatric surgery
15. Weight loss > 5% in the past 1 month
16. Metallic implants (including incompatible pacemakers, AICD, metallic heart valves) or other contraindications to MRI
17. Claustrophobia
18. Any factors likely to limit adherence to study protocol (e.g., dementia; alcohol or substance abuse; history of unreliability in medication taking or appointment keeping; significant concerns about participation in the study from spouse, significant other, or family members)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Changes in hepatic Magnetic Resonance Imaging-Proton Density Fat Fraction and concentrations of acylglycines, glutathione, cytokines, oxidative stress markers, and 1-carbon cycle metabolites from baseline to 26 weeks | From the initiation to end of the treatment at 26 weeks
Differences in concentrations of acylglycines, glutathione, cytokines, oxidative stress markers, and 1-carbon cycle metabolites between subjects with MASLD and controls | From enrollment to the completion of baseline metabolic assessment (within 8 weeks)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Time Frame: Beginning 3 months and ending 3 years after the publication of results